CLINICAL TRIAL: NCT05209607
Title: A Multicenter Open-label Randomized Controlled Trial of Social Media-based Bundle Care in Patients With Exacerbation of Chronic Obstructive Pulmonary Disease.
Brief Title: Social Media-based Bundle Care of AECOPD Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Peking University (Other); Xuanwu Hospital, Beijing (Other); Beijing Anzhen Hospital (Other); Beijing Tongren Hospital (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Emergency General Hospital (Other); Beijing Jishuitan Hospital (Other); Beijing Luhe Hospital (Other); Beijing Shijingshan Hospital (Unknown); Beijing Jingmei Group Hospital (Unknown)
Responsible Party: Principal Investigator, Yingxiang Lin, Chief physician of Department of Respiratory and Critical Care Medicine, Beijing Institute of Respiratory Medicine, Beijing Chao-Yang Hospital, Capital Medical University,, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Z201100005520031
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Acute Exacerbation of COPD; Pulmonary Disease, Chronic Obstructive; COPD; Lung Diseases, Obstructive; Readmission Rate; Mobile Medical; Bundle Care; Mobile Telemedicine
Keywords: Readmission rate; Chronic Obstructive Pulmonary Disease; Randomized Controlled Trial; Bundle care; Mobile Telemedicine; Mobile medical; Acute Exacerbation of Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Participants will be given mobile medical and bundle care
  Interventions: Other: Mobile Medical and bundle management
- Control group (Other): Participants will be given mobile medical and standard of care.
  Interventions: Other: Mobile Medical and standard of care

INTERVENTIONS:
Other: Mobile Medical and bundle management — Based on the current follow-up management platform of respiratory disease, the WeChat official account will be designed and used to provide health education for patients, such as smoking cessation, reasonable diet, appropriate exercise, etc., and monitor some physiological indicators (such as body temperature, weight, the score of mMRC, etc.) and guide patients to standardize medication and pulmonary rehabilitation.
  Arms: Interventional group
Other: Mobile Medical and standard of care — Based on the mobile medical, participants will receive advice on standard medication only.
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease(COPD) is an incompletely reversible and progressive pulmonary disease characterized by airflow restriction, which is the third leading cause of death worldwide, accounting for 6% of all deaths worldwide. Acute exacerbation (AE) of COPD can accelerate the decline of lung function, worsening pulmonary symptoms, and increase the risk of death in patients. Health education, inhaled technical guidance training, individual self-management, psychological counseling, home oxygen therapy, nutritional support, and other comprehensive interventions can help improve the lung function of COPD patients, alleviate clinical symptoms, improve the quality of life. While a number of COPD applications have been developed, few provide comprehensive assessment and guidance for these kinds of patients. Therefore, the investigators aim to establish a bundle care mode based on the mode of "hospital-home-community-patient", clarify the impact of the management on prognosis, and evaluate the effect of mobile medical-assisted bundle management mode. In this randomized controlled trial(RCT), AECOPD patients will be divided into interventional or control groups randomly. Patients in the interventional group will receive mobile medication and standard of care at the same time (bundle care mode). While patients in the control group will receive standard of care only (traditional management mode). This study will be conducted to compare the effects of traditional and bundle care modes, and to formulate the implementation path and specifications of bundle care for AECOPD patients after discharge in China.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD Patients with pulmonary function grade GOLD2-4;
* Aged between 45 and 70 years old;
* Have a smartphone, and can skillfully use mobile Wechat official account;
* Willing to use Wechat official accounts to manage COPD;
* Willing to accept outpatient follow-up;
* Signed informed consent.

Exclusion Criteria:

* Patients with asthma, bronchiectasis, tuberculosis, or other diseases;
* Patients with malignant tumors, liver and kidney failure, limb dyskinesia, and other diseases;
* Unstable angina pectoris in recent one month, myocardial infarction within a half year, severe arrhythmia, uncontrollable congestive heart failure, or poor blood pressure control (systolic blood pressure > 140mmHg and/or diastolic blood pressure > 90mmHg);
* Cognitive impairment;
* Combined with respiratory failure;
* With a life expectancy of less than one year;
* Plan to or participating in a COPD management project or mobile Wechat official account project;
* Completed another trial within 30 days.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Readmission rate due to acute exacerbation of COPD within one year | One year
  Collected within one year after discharge

SECONDARY OUTCOMES:
The time interval from discharge to the next acute exacerbation of COPD | One year
  Collected within one year after discharge
The times of acute exacerbation of COPD | One year
  Collected within one year after discharge
The score of subjective symptom | One year
  Collected within one year after discharge. We will use modified Medical Research Council (mMRC) Dyspnoea Scale, COPD Assessment Test (CAT), St. George's Respiratory Questionnaire (SGRQ),Hospital Anxiety and Depression Scale (HADS) and Borg scale to assecc.
The changes of spirometry | One year
  Collected within one year after discharge. FEV1/FEV, FEV1 %pre，FVC, DLCO and RV/TLC etc will be collected.
The changes of arterial blood gas analysis | One year
  Collected within one year after discharge. PaO2, PaCO2, BE, HCO3-, Lac, K+, Na+, Glu etc will be collected.
The changes of percent of eosinophil count | One year
  Collected within one year after discharge
Average annual medical cost | One year
  Collected within one year after discharge
The types and proportions of adverse events occurred during using WeChat official account. | One year
  Collected within one year after discharge
Compliance index | One year
  It includes drug treatment compliance, mastery of drug inhalation skills, smoking cessation, improvement of nutritional status, changes of mental health status, compliance and mastery of lung rehabilitation exercise, and patients' cognitive level of chronic obstructive pulmonary disease.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothnie KJ, Mullerova H, Smeeth L, Quint JK. Natural History of Chronic Obstructive Pulmonary Disease Exacerbations in a General Practice-based Population with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2018 Aug 15;198(4):464-471. doi: 10.1164/rccm.201710-2029OC. PMID 29474094
- [Background] Sobnath DD, Philip N, Kayyali R, Nabhani-Gebara S, Pierscionek B, Vaes AW, Spruit MA, Kaimakamis E. Features of a Mobile Support App for Patients With Chronic Obstructive Pulmonary Disease: Literature Review and Current Applications. JMIR Mhealth Uhealth. 2017 Feb 20;5(2):e17. doi: 10.2196/mhealth.4951. PMID 28219878